CLINICAL TRIAL: NCT01978743
Title: Advanced Neuroimaging Evaluation of the Central Nervous System Biological Changes Associated With Efavirenz Therapy Switch to an Raltegravir-based Regimen
Brief Title: Advanced Neuroimaging Evaluation of CNS Changes Associated With Efavirenz Therapy Switch to an Raltegravir-based Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Nina Lin, MD, Assistant Professor in Medicine, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NeuroHIV002
Record Dates: First submitted 2013-10-20; First posted 2013-11-07 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: HIV; HIV-associated Neurocognitive Disorder; Neurotoxicity
Keywords: HIV; HIV-associated neurocognitive disorder; neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Raltegravir Potassium; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (Experimental): Switch from Atripla (EFV/FTC/TDF) to raltegravir (RAL) + Truvada (FTC/TDF). Raltegravir will be administered 400mg twice-a-day with Truvada for 8 weeks.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Switch from Atripla to Raltegravir 400mg BID + Truvada (FTC/TDF) for total of 8 weeks
  Other Names: Raltegravir (Isentress) 400mg BID

SUMMARY:
In this study investigators will use a multi-modal imaging approach of MRS and fMRI to comprehensively assess the biological changes in the brain associated with EFV-based regimen (EFV/FTC/TDF), specifically alterations in the brain circuitry, function and local neurochemistry, and their correlation with neuropsychological function.

DETAILED DESCRIPTION:
In a cohort of HIV-infected patients who are clinically stable on the commonly use regimen of EFV/emtricitabine (FTC)/truvada (TDF) or Atripla, investigators propose to replace the EFV component with an integrase inhibitor, Raltegravir (RAL), given as the RAL and FTC/TDF to evaluate the EFV-related neural alterations. This is a multidisciplinary study which will be lead by Dr. Nina Lin, in collaboration with the research teams of Dr. Alexander Lin, Director of the Center for Clinical Spectroscopy, and Dr. Emily Stern, Director of the Functional Neuroimaging Laboratory, both members of the Brigham and Women's Department of Radiology at Harvard Medical School, as well as Dr. Jane Epstein, a researcher in Dr. Stern's research group. Dr. Epstein is a staff psychiatrist at Brigham and Women's hospital with extensive experience and expertise in research on abnormalities of affective and motivational processing in the context of neuropsychiatric disorders. Investigators will utilize the established clinical research platform in the Infectious Disease outpatient clinical practice at the Brigham and Women's Hospital, where there is currently have many ongoing HIV-related studies and a large panel of HIV-infected patients motivated to be involved in clinically relevant research. Investigators propose to use advanced neuroimaging to measure biologically changes in the brain associated with long-term EFV use with the following specific aims:

1. Determine changes in neurometabolites measured by MRS in the brain associated with long-term EFV use
2. Assess for alterations in neural activity correlated with affective symptoms associated with EFV vs RAL use using fMRI, and their associations with changes in neurometabolites assessed by MRS, and with changes in cognition assessed by Trail Making and Digit Substitution Tests.
3. Determine changes in emotion, cognition and sleep quality after switching from EFV to RAL, and how they correlate with subject treatment preference.

This clinical study will extend our current understanding of EFV neurotoxicity by further defining the nature of these biological changes. Further elucidation of the neurobiological underpinnings of EFV-induced CNS toxicity will have clinical relevance in improving the quality of life and drug adherence of HIV-infected patients on ART, especially among older patients or those with baseline neuropsychiatric disorders, whom at baseline are more vulnerable to neurocognitive decline from long-term HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HIV-infected individuals on suppressive regimen with EFV/FTC/TDF, for at least 6 months
2. Undetectable HIV-1 RNA virus load for at least 6 months
3. No co-infections with active hepatitis B and C
4. Presence of at least moderate symptoms on 2 out of 3 subcores on the DASS
5. No known active HIV-related and non-HIV related CNS infections
6. Estimated glomerular filtration rate (EGFR) >60 ml/min
7. Consent to switching to EVG/COBI/FTC/TDF
8. Ages 18 - 65

Exclusion Criteria:

1. History of CNS opportunistic infections or active CNS infections
2. History of severe psychiatric disorder (excluding depression and anxiety)
3. History of chronic neurological disorders, such as epilepsy or multiple sclerosis
4. History of or current significant substance abuse or dependence and/or heavy alcohol use (>12 oz/wk)
5. Any women who may be pregnant (positive urine pregnancy test or unprotected sex in 2 weeks prior to scan) or known to be pregnant
6. Contraindications to undergoing fMRI, including metallic implants, claustrophobia, and medical conditions or medications that significantly affect cerebral blood flow or function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: All participants are switched from Atripla (EFV/FTC/TDF) to raltegravir (RAL) + truvada (FTC/TDF).
  Raltegravir will be administered 400mg twice-a-day.
Period: Overall Study
Arm/Group | Raltegravir
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Raltegravir: All 10 participants were switched from Atripla to twice daily Raltegravir and Truvada (FTC/TDF)
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Neurometabolites Based on Magnetic Resonance Spectroscopy (MRS)
Description: Assess the levels of neuro-metabolites measured by MRS at week 0 before switching to the efavirenz-based therapy. Two areas of the brain: 1) posterior cingulate gyrus and 2) anterior cingulate will be assessed for the levels of brain creatine (Cr), gamma-aminobutyric acid (GABA) and glutathione (GLU).
Time Frame: week 0 and week 8
Population: The arbitrary units are expressed as the output from MRS software. While similar to concentration (mM) due to assumptions in the software, it is best expressed as arbitrary units for comparison from week 0 to week 8.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Raltegravir: Switch from Atripla (EFV/FTC/TDF) to raltegravir (RAL) + Truvada (FTC/TDF). Raltegravir will be administered 400mg twice-a-day with Truvada for 8 weeks.
  Drug switch from Atripla: Switch from Atripla to Raltegravir 400mg BID + Truvada (FTC/TDF) for total of 8 weeks
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
arbitrary units
  Pre-switch Posterior Cingulate Creatine | 19.38 (1.82)
  Post-switch Posterior Cingulate Creatine | 18.94 (4.01)
  Pre-switch Posterior Cingulate Glutamate | 27.83 (5.06)
  Post-switch Posterior Cingulate Glutamate | 24.95 (4.54)
  Pre-switch Posterior Cingulate GABA | 5.27 (0.74)
  Post-switch Posterior Cingulate GABA | 5.32 (1.85)
  Pre-switch Anterior Cingulate Creatine | 14.86 (2.18)
  Post-switch Anterior Cingulate Creatine | 14.34 (2.92)
  Pre-switch Anterior Cingulate Glutamate | 19.09 (3.83)
  Post-switch Anterior Cingulate Glutamate | 22.25 (6.21)
  Pre-switch Anterior Cingulate GABA | 4.73 (1.55)
  Post-switch Anterior Cingulate GABA | 3.14 (2.12)

2. Primary Outcome: Neural Activation Networks Using Functional Magnetic Resonance Imaging (fMRI)
Description: Assess changes in neural activation correlated with affective disturbances associated with EFV vs. RAL using fMRI employing a paradigm that probes affective symptomatologies typical with EFV use; anxiety/dysphoria and affective dysregulation, and their association with changes in cognitive function. Four brain regions of interests (ROIs) are specified to show the differential frontal-limbic activation patterns in the task-evoked neural responses to the 3 linear contrasts of Pre-/Post-/ Pre-vs. Post-switch: [Negative Word vs. Neutral Word] x [No-Go Trial Block vs. Go Trial Block]: anterior Frontal Pole (aFP), posterior Cingulate Gyrus (pCG), dorsal anterior Cingulate Gyrus (daCG), Left Hippocampus (LHC). A linear mixed-effects model is utilized to examine the effect sizes of the key Regimen/Condition contrasts, with the Subject factor as the random-effect, and Age incorporated as a co-variate of no interest. A z-score is the Mean with a SD=1 and Measure of Dispersion equal to 1.
Time Frame: week 0 and week 8
Population: 8 of 10 enrolled patients passed QA testing to qualify for final fMRI data analyses. The 3 linear contrasts of Pre-switch/Post-switch/Pre- vs. Post-switch: [Neg vs.Neu] x [No-Go vs. Go] are reported as z-score (standardized effect size measures with SD=1). Z-score is obtained for each subject, group Z-score is obtained via a mixed-effects model.
Measure: Number; unit: z-score
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
z-score
  PreVsPostXNegVsNeuXNoGoVsGo: aFP | 3.19
  PreVsPostXNegVsNeuXNoGoVsGo: pCG | 3.00
  PreVsPostXNegVsNeuXNoGoVsGo: daCG | -2.53
  PreVsPostXNegVsNeuXNoGoVsGo:LHC | -3.64
  Pre: NegVsNeuXNoGoVsGo: aFP | 4.01
  Pre: NegVsNeuXNoGoVsGo:pCG | 3.61
  Pre: NegVsNeuXNoGoVsGo: daCG | -2.94
  Pre: NegVsNeuXNoGoVsGo: LHC | -3.07
  Post: NegVsNeuXNoGoVsGo: aFP | -3.03
  Post: NegVsNeuXNoGoVsGo: pCG | -3.13
  Post: NegVsNeuXNoGoVsGo: daCG | 3.65
  Post: NegVsNeuXNoGoVsGo: LHC | 2.88

3. Secondary Outcome: Other Neurometabolite Changes Measured by MRS
Description: Use MRS to evaluate a fuller panel of known neurometabolites (in addition to the primary endpoints) to evaluate for prominent and significant changes associated with EFV use.
Time Frame: week 0 and week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
arbitrary units
  Pre-switch Posterior Cingulate Glutathione | 5.11 (1.18)
  Post-switch Posterior Cingulate Glutathione | 4.70 (1.51)
  Pre-switch Posterior Cingulate Aspartate | 4.32 (0.95)
  Post-switch Posterior Cingulate Aspartate | 3.31 (0.97)
  Pre-switch Anterior Cingulate Glutathione | 4.25 (1.01)
  Post-switch Anterior Cingulate Glutathione | 3.18 (1.08)
  Pre-switch Anterior Cingulate Aspartate | 3.15 (1.28)
  Post-switch Anterior Cingulate Aspartate | 2.18 (1.61)

4. Secondary Outcome: Neurocognitive Changes Measured by a Panel of Indexes: WAIS-R, HAMD, DASS-21, FRSBE, STAI
Description: Assess for changes in cognitive and affective function prior to and after switching off EFV-based regimen. Indexes used to access neurocognitive changes included:
  1. Wechsler Adult Intelligence Scale (WAIS-R) Digital Symbol Substitution Test: sensitive to brain dmamage, dementia, age and depressive changes. Range of 0-100, the higher the score the better the person's performance
  2. Hamilton Rating Scale for Depression (HAMD): Measure of depression. Score of 0-7 is normal, score of >20 is moderate/severe depression
  3. Depression Anxiety Stress Scale (DASS-21) the lower the score, the less severe depression, anxiety and stress. Scale range of 0-63
  4. Frontal Systems Behavior Scale (FRSBE): Increased score indicates greater behavioral impairment associated with frontal systems, range 37.2 to 186
  5. Spielberger state trait anxiety inventory (STAI): the higher the score the greater then anxiety level, range of 20 to 80.
Time Frame: week 0 and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
units on a scale
  pre-switch WAIS | 48.1 (12.53838551)
  post-switch WAIS | 53.5 (12.00231459)
  pre-switch FRSBE | 79.2 (13.07074766)
  post-switch FRSBE | 72.4 (9.834180754)
  pre-switch HAMD | 4.7 (3.860051813)
  post-switch HAMD | 2.7 (3.020301677)
  pre-switch DASS depression | 6.4 (9.834180754)
  post-switch DASS depression | 3.4 (3.777124126)
  pre-switch STAI | 29.4 (5.481281278)
  post-switch STAI | 27.2 (6.528569692)

5. Secondary Outcome: Fasting Lipid Profile
Description: Measure the change in fasting lipid panel prior to and after switching off EFV-based regimen.
Time Frame: week 0 and week 8
Population: Change in lipid panel pre- and post-switch to RAL-based regimen
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
mg/dL
  pre-switch total cholesterol | 200.9 (37.02)
  post-switch total cholesterol | 176.7 (26.20)
  pre-switch HDL | 58.8 (9.69)
  post-switch HDL | 53.1 (13.42)
  pre-switch LDL | 118.8 (31.56)
  post-switch LDL | 103.5 (24.08)
  pre-switch triglyceride | 116.4 (69.62)
  post-switch triglyceride | 100.6 (54.52)

6. Secondary Outcome: Sleep Quality
Description: Assess for changes in sleep pattern and quality prior to and after switching off EFV-based regimen through a self-administered Pittsburg Sleep Quality Index (PSQI). Measure consists of 19 items with each weighted on 0-3 scale and the sum produces a total score, which ranges from 0-21. The lower the score the healthier the sleep quality.
Time Frame: week 0 and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
units on a scale
  pre-switch PSQI index | 5.3 (3.06)
  post-switch PSQI index | 3.8 (1.99)

7. Secondary Outcome: ART Regimen Preference
Description: Evaluate patient preference in ART regimen (Atripla, EFV/FTC/TDF versus RAL + FTC/TDF) through self-administered questionnaires.
Time Frame: week 0 and week 8
Population: Each participant was asked a single self-administered question on their ART preference and asked to chose one of the 3 answers; 1. prefer to take Atripla, 2. prefer RAL-based regimen (that they received in study) or 3. no preference.
Measure: Number; unit: participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
participants
  Prefer Raltegravir-based ART | 7
  Prefer Atripla (EFV-based ART) | 0
  No preference | 3

8. Secondary Outcome: Markers of Immune Activation
Description: Change in markers of immune activation and inflammation associated with change to RAL (ie, sCD14, IL-6, hsCRP, D-dimer, CRP, LPS, sCD163, EndoCab)
Time Frame: week 0 and week 8
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
pg/ml
  pre-switch sCD14 | 3652333.6 (771769.196)
  post-switch sCD14 | 3135828.52 (791445.1417)
  pre-switch IP-10 | 195.84 (74.57)
  post-switch IP-10 | 202.85 (55.58)
  pre-switch sCD163 | 672844 (281620)
  post-switch sCD163 | 733536 (378.958)
  pre-switch MCP-1 | 95.578 (34.14)
  post-switch MCP-1 | 92.794 (56.25)
  pre-switch IL-6 | 1.49 (0.68)
  post-switch IL-6 | 1.69 (0.89)
  pre-switch TNFR1 | 771.18 (145.46)
  post-switch TNFR1 | 829.12 (130.66)

9. Secondary Outcome: Change in Level of EFV and Metabolites
Description: Correlate change in level of EFV and metabolites with neurocognitive and neuroimaging changes
Time Frame: week 0 and week 8
Population: Level of EFV (efavirenz) in Atripla and its two known metabolites known to cause cerebral side effects, 7-hydroxy (OH) EFV and 8-OH EFV, were measured in the plasma prior to switch off Atripla and after 8 weeks of RAL-based regimen (no EFV).
Measure: Number; unit: participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
participants
  pre-switch detectable 7-OH and 8-OH EFV metablites | 9
  post-switch detectable 7-OH and 8-OH EFVmetaboites | 1

ADVERSE EVENTS:
Arm/Group | Raltegravir
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No